CLINICAL TRIAL: NCT07331506
Title: Validation of the Oncoliq Test for the Early Detection of Breast Cancer.
Status: Recruiting | Type: Observational
Sponsor: Oncoliq US Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: DIM001
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer Detection; Breast Cancer Early Stage Breast Cancer (Stage 1-3); Breast Cancer Female; Breast Cancer - Ductal Carcinoma in Situ (DCIS); Breast Cancer - Infiltrating Ductal Carcinoma; Breast Cancer With Low to Intermediate HER2 Expression; Breast Cancer (Early Breast Cancer); Breast Cancer - Female
Keywords: Breast cancer; Detection; Liquid biopsy; miRNAs
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected and processed to obtain plasma, which will be stored for future analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast Cancer Cohort: Participants with a confirmed diagnosis of breast cancer, prior to surgery or systemic treatment.
  Interventions: Other: Peripheral blood draw
- Healthy Control Cohort: Cancer-free volunteers confirmed by breast imaging (BI-RADS 1 or 2) and without a prior history of cancer.
  Interventions: Other: Peripheral blood draw

INTERVENTIONS:
Other: Peripheral blood draw — Collection of a blood sample for plasma isolation and miRNA analysis.

SUMMARY:
Cancer continues to be one of the most significant public health issues worldwide. Thanks to early detection, the mortality rate of certain types of cancer has decreased significantly. However, the lack of accessible, low-cost, non-invasive, non-toxic, and easy-to-implement diagnostic methods results in late diagnoses, leading to 1 in every 6 people dying from cancer today.

MicroRNAs (miRNAs) are small non-coding RNAs that regulate gene expression and are found both inside cells and in bodily fluids such as blood and urine. Several studies have demonstrated their role in human diseases, especially cancer, where tumors release miRNAs into the bloodstream that can be used as biomarkers for early detection.

The research and development team at Oncoliq SAS identified a panel of miRNAs associated with breast cancer, with a detection performance of 82% sensitivity and 83% specificity, validated in exploratory and preliminary confirmatory studies. These results led to the filing of a patent based on liquid biopsy technology.

The objective of this protocol is to establish a panel of miRNAs for the early detection of breast cancer using samples from breast cancer patients and a cancer-free control group. Validation of the miRNAs will be carried out through RT-qPCR. This stage constitutes the analytical validation of the biomarkers, with the goal of developing an algorithm capable of classifying individuals with and without breast cancer. In future stages, a pilot clinical trial is planned to evaluate test implementation and clinical validation.

ELIGIBILITY:
Inclusion Criteria:

Group 1 - Breast Cancer:

Age between 40 and 70 years Diagnosis of breast cancer at any stage No prior surgical treatment No prior antineoplastic treatment Pathology report available at the time of enrollment Signed informed consent

Group 2 - No Cancer (Control):

Age between 50 and 70 years No diagnosis or personal history of any type of cancer Digital mammography and breast ultrasound showing no breast pathology (BI-RADS 1 or 2) Signed informed consent

Exclusion Criteria:

Refusal to sign the informed consent Communication issues that hinder understanding (hearing loss, blindness, intellectual disability, or dementia) Venipuncture for blood collection impracticable or posing a risk Personal history of previous cancer

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: The study population consists of two groups of female participants. Group 1 (Breast Cancer): Women aged 40-70 years with a confirmed diagnosis of breast cancer at any stage, prior to any surgical or antineoplastic treatment, and with a pathology report available at enrollment.
  Group 2 (Control - No Cancer): Women aged 50-70 years with no current or past history of cancer and normal breast imaging findings (digital mammography and breast ultrasound, Bi-RADS 1/2).
  All participants must be able to provide written informed consent. Exclusion criteria include inability to understand the study procedures, medical conditions that make venipuncture unsafe or unfeasible, and any prior history of cancer.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Enrollment of 300 Participants | October to December 2025
  Successful recruitment and enrollment of a total of 300 eligible participants across both study groups within the planned recruitment period.

SECONDARY OUTCOMES:
Development of a Machine Learning Classification Algorithm | December 2025 to March 2026
  Creation and validation of a machine learning model capable of distinguishing between individuals with breast cancer and cancer-free controls based on blood-derived biomarkers.

CONTACTS AND LOCATIONS:
Locations (1):
- DIM Centros de Salud, Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: 'Breast Cancer Diagnostic and Treatment' — https://patentscope.wipo.int/search/en/detail.jsf?docId=WO2023170659